CLINICAL TRIAL: NCT05343533
Title: Impact of Probiotic Administration on Mood, Psychological Traits, Physical Activity, Stress, and Sleep Quality
Brief Title: Probiotic Administration on Mood
Acronym: PAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Collaborators: Increnovo, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-19-212
Record Dates: First submitted 2022-03-29; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Depression; Sleep; Stress; Anxiety; Mood Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Mood Disorders | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: andomized, double-blind, placebo-controlled, parallel study design that will evaluate the ability of a probiotic to influence mood, depressive symptoms, anxiety, sleep quality, and other personality traits in a group of healthy men and women
Who Masked: Participant, Investigator
Masking Description: All supplements were blinded from participant and investigator by a third party
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Probiotic (Experimental): A mixture of probiotic strains (2.5 gram daily doses of 4 x 109 CFU/packet) of the following species (Lactobacillus fermentum, Lactobacillus rhamnosus, Lactobacillus plantarum, Bifidobacterium longum).
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Maltodextrin capsule
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — After baseline or initial testing, participants will be randomly assigned in a double-blind fashion to ingest on a daily basis for 6 weeks either a placebo or a probiotic supplement. Identical follow-up measurements will then occur each visit after taking their assigned supplement. After 6 weeks of administration, the supplementation protocol will stop and a final evaluation will be completed 3 weeks later (9 weeks after initial administration) to assess any residual impact of the assigned supplement after a 3-week washout.

SUMMARY:
Researchers are looking to examine the impact of probiotic administration on symptoms commonly associated with depression, anxiety, stress, sleep quality, and associated emotional responses in healthy men and women.

DETAILED DESCRIPTION:
In recent years, the presence and awareness of a connection between the intestines and the brain has expanded leading to the understanding of developed communication pathways between the nervous, endocrine, and immune systems. Intestinal bacterial flora are active contributors to this axis through cellular signaling pathways and the release of immune system components, which fundamentally impact the function and action of various physiological systems. Interest in this area evolved through the understanding that various microbiota can produce neuroactive substances and neurotransmitters involved with the endocrine and autonomic nervous system pathways. This research has expanded to state that various bacterial products can influence cognitive functions, involving types of memory and problem-solving. Recent findings have begun to report on the impact that probiotic administration may have on mood, anxiety, and depression. Finally, recent work by Marotta et al. provided some of the first preliminary evidence that probiotic use may also impact mood and sleep quality. While initial work has developed this foundation, very little controlled research is available to help understand key contributing factors. For example, many key questions remain that future research should address to help better understand any impact probiotics may have on mood, depression, and anxiety. Some of these questions include:

Do all forms (genus, strain, etc.) of probiotics exert these impacts? How quickly do they exert impact? How large is the impact? Are certain aspect of affect more impacted than others? Once supplemented, how long is the residual impact (if there is any)? To help provided more guidance towards some of these basic research questions, this study is being proposed. The purpose of the study is to expand upon the previous work of Marotta et al. and determine the impact of probiotic administration on mood, depressive symptoms, anxiety, sleep quality, and other personality traits in a larger group of healthy men and women. This study will expand on the supplementation regimen and include a wider variety of hormonal assessments than what has previously been completed using this combination of probiotics.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 - 50 years
* has a body mass index between 18.5 - 30 kg/m2.
* Anyone with a body mass index between 30 - 32 kg/m2, but has a body composition <25% fat -for men and <35% for women will be accepted into the study
* has been weight stable for the past three months (defined as less than a 5% variation in body -mass over this time)
* is determined to be healthy through completion of a health history questionnaire

Exclusion Criteria:

* Are currently diagnosed or being treated for any cardiac, respiratory, endocrine, psychiatric, musculoskeletal, - renal, hepatic, neuromuscular or metabolic disease or disorder that in the judgement of the study participant's personal physician or research nurse that will preclude their safe participation or will contraindicate quality control over the collected data
* are currently diagnosed with or are being treated for celiac disease, lactose intolerance, digestive insufficiencies or other gastrointestinal complications such as irritable bowel syndrome, ulcerative colitis, etc.
* report having used anabolic steroids within the past 30 days
* report have used any illicit or recreational drugs within the past 30 days
* report the intake of any prescription or over-the-counter medications (i.e., antibiotics) that may impact study outcomes
* report the current use of any dietary supplements known to impact digestion or sleep quality for the past 30 days
* report already taking a probiotic within the past 30 days
* have been actively trying to lose weight
* are currently following a ketogenic or low carbohydrate diet within the past 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Index II | 6 Weeks
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.
  Total Score Levels of Depression 0-10 = These ups and downs are considered normal 11-16 = Mild mood disturbance 17-20 = Borderline clinical depression 21-30 = Moderate depression 31-40 = Severe depression over 40 = Extreme depression
COPE Inventory | 6 weeks
  The COPE Inventory is a multidimensional coping inventory to assess the different ways in which people respond to stress. Five scales (of four items each) measure conceptually distinct aspects of problem-focused coping (active coping, planning, suppression of competing activities, restraint coping, seeking of instrumental social support); five scales measure aspects of what might be viewed as emotion-focused coping (seeking of emotional social support, positive reinterpretation, acceptance, denial, turning to religion); and three scales measuring coping responses that arguably are less useful (focus on and venting of emotions, behavioral disengagement, mental disengagement).
Leiden Index of Depression Sensitivity - Revised | 6 weeks
  The Leiden Index of Depression Sensitivity (LEIDS) measures cognitive reactivity (CR) to sadness, an aspect of cognitive vulnerability to depression, conceptually similar to rumination. A higher total score on all the subscales except acceptance and coping shows higher CR.
Pittsburgh Sleep Quality Index | 6 weeks
  A self-rated questionnaire to assess sleep quality and disturbances
  19 self-reported items Minimum score: 0; Maximum score: 21 Higher scoring indicated worse sleep quality
State-Trait Anxiety Inventory form Y1 and Y2 | 6 weeks
  Measure of trait and state anxiety. All items on the scale are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety. The STAI is appropriate for those who have at least a sixth-grade reading level.
Behavioral Avoidance/Inhibition Scale | 6 weeks
  A measure of motivation to approach goal-oriented outcomes. Higher scores correspond to higher motivation to avoid goal oriented outcomes, lower scores indicate lower motivation to avoid goal-oriented outcomes.
Bowel Health Questionnaire | 6 weeks
  Measure of bowel health. Lower scores indicate lower number of GI disturbances and higher scores indicate higher number of GI disturbances

SECONDARY OUTCOMES:
Hours Asleep | 6 weeks
  Total hours asleep each night as obtained through a fit bit activity monitor
Minutes Awake | 6 weeks
  Total minutes awake each night as obtained through a fit bit activity monitor
Number of awakenings | 6 weeks
  Number of times awakened each night as obtained through a FitBit activity monitor
Minutes of restlessness | 6 weeks
  Total minutes of restlessness each night as obtained through a FitBit activity monitor
Number of times Restless | 6 weeks
  Number of times restless each night as obtained through a FitBit activity monitor
Total time Awake and Restless | 6 weeks
  Total minutes of time awake and restless each night as obtained through a FitBit activity monitor
Total time in Bed | 6 weeks
  Total time in bed each night as obtained through a FitBit activity monitor
Calories Burned | 6 weeks
  Total KCal burned on average each day as obtained through a FitBit activity monitor
Steps | 6 weeks
  Total number of steps on average each day as obtained through a FitBit activity monitor
Distance | 6 weeks
  Total distance traveled each day on average each day as obtained through a FitBit activity monitor
Minutes Sedentary | 6 weeks
  Total minutes sedentary on average each day as obtained through a FitBit activity monitor
Minutes Lightly Active | 6 weeks
  Total minutes Lightly active on average each day as obtained through a FitBit activity monitor
Minutes Fairly Active | 6 weeks
  Total minutes Fairly active on average each day as obtained through a FitBit activity monitor
Minutes Very Active | 6 weeks
  Total minutes Very active on average each day as obtained through a FitBit activity monitor
Active Calories | 6 weeks
  Total minutes of active calories expended on average each day as obtained through a FitBit activity monitor
Body Composition | 6 weeks
  DEXA derived fat mass and fat free mass and bodyfat percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Lindenwood University, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerksick CM, Moon JM, Walden KE, Hagele AM, Allen LE, Gaige CJ, Krieger JM, Jager R, Pane M, Mumford P. Multi-strain probiotic improves subjective sleep quality with no impact on body composition, hemodynamics, and physical activity. Benef Microbes. 2024 Jan 31;15(2):179-194. doi: 10.1163/18762891-bja00002. PMID 38350465
- [Derived] Walden KE, Moon JM, Hagele AM, Allen LE, Gaige CJ, Krieger JM, Jager R, Mumford PW, Pane M, Kerksick CM. A randomized controlled trial to examine the impact of a multi-strain probiotic on self-reported indicators of depression, anxiety, mood, and associated biomarkers. Front Nutr. 2023 Aug 31;10:1219313. doi: 10.3389/fnut.2023.1219313. eCollection 2023. PMID 37720373